CLINICAL TRIAL: NCT03562260
Title: Result of Bipolar Surgical Release in Congenital Muscular Torticollis
Brief Title: Bipolar Surgical Release in Congenital Muscular Torticollis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: si049/2013
Record Dates: First submitted 2018-05-21; First posted 2018-06-19 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Congenital Muscular Torticollis
MeSH Terms: conditions — Congenital torticollis

STUDY DESIGN:
Intervention Model Description: only 1 group in children who received the bipolar release
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children who had bipolar release (Experimental): children who had bipolar release are included
  Interventions: Procedure: bipolar release

INTERVENTIONS:
Procedure: bipolar release — the bipolar release is the surgery that cut the origin and insertion of the sternocleidomastoid muscle that cause the torticollis from its contracture

SUMMARY:
The congenital muscular torticollis is common disease in children.The indication for surgery is the children have persist deformity after 1 year old.Many surgical treatment had proposed such as unipolar release and bipolar release.By author experience the bipolar release had better results from complete cut the muscle both origin and insertion.This study wants to study the results of treatment in term of recurrence of the deformity.

DETAILED DESCRIPTION:
the study perform in children with congenital muscular torticollis

ELIGIBILITY:
Inclusion Criteria:

* 1. all children age ranged from 5-15 years old who received the surgical treatment by bipolar release in the hospital.

Exclusion Criteria:

* 1. no history of surgery at the neck 2. no history of congenital anomalies and syndrome that effect the neck

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2019-08-09 (Estimated); Study Completion 2019-08-09 (Estimated)

PRIMARY OUTCOMES:
ImageJ scoring system | no torticollis after 1 year of surgery
  measurement from pictures of head and face compared to normal children score 1-3 in 5 measurement in total score of 15 as interval scale score has 4 grade 13-15 is excellent results score 10-12 good result 7-9 fair less than 6 score is poor result after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Kamolporn Kaewpornsawan, Principal Investigator — Department of Orthopaedic Surgery,Faculty of Medicine,Siriraj Hospital,Mahidol University,Bangkok,Thailand
Locations (1):
- Prof.Dr.Kamolporn Kaewpornsawan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
no sharing IPD data

REFERENCES:
- [Background] Lee EH, Kang YK, Bose K. Surgical correction of muscular torticollis in the older child. J Pediatr Orthop. 1986 Sep-Oct;6(5):585-9. doi: 10.1097/01241398-198609000-00011. PMID 3760169
- [Background] Sudesh P, Bali K, Mootha AK, Dhillon MS. Results of bipolar release in the treatment of congenital muscular torticolis in patients older than 10 years of age. J Child Orthop. 2010 Jun;4(3):227-32. doi: 10.1007/s11832-010-0254-x. Epub 2010 Mar 26. PMID 21629376
- [Background] Shim JS, Jang HP. Operative treatment of congenital torticollis. J Bone Joint Surg Br. 2008 Jul;90(7):934-9. doi: 10.1302/0301-620X.90B7.20339. PMID 18591606